CLINICAL TRIAL: NCT00889109
Title: Proprioception of the Glenohumeral Joint Following Open and Arthroscopic Repair for Anterior Shoulder Instability
Brief Title: Shoulder Proprioception Following Open and Arthroscopic Instability Repair
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Ariel Oran M.D, The Shoulder Surgery Unit, Sheba Medical Center, Tel Hashomer, Israel
Other Study IDs: SHEBA-09-7068-AO-CTIL
Record Dates: First submitted 2009-04-26; First posted 2009-04-28 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Shoulder Proprioception; Open Capsular Shift; Arthroscopic Bankart Repair; Unrestricted Arm Movement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Open Capsular Shift
  Interventions: Other: Three dimensional unrestricted arm movements
- 2: Arthroscopic Bankart Repair
  Interventions: Other: Three dimensional unrestricted arm movements
- 3: Healthy controls
  Interventions: Other: Three dimensional unrestricted arm movements

INTERVENTIONS:
Other: Three dimensional unrestricted arm movements — The subjects will carry out three dimensional unrestricted arm movements. The subjects' movements will be recorded by optoelectronic infrared cameras and software. Assessment of smoothness parameters of subjects' movements will allow discriminating between subjects with intact or impaired proprioception.

SUMMARY:
Shoulder dislocations are common and may result in functionally disabling instability. Disruption of the shoulder capsuloligamentous complex during shoulder dislocation is related to poor proprioceptive and stabilizing capabilities of the joint. It has been demonstrated that surgical restoration of the normal glenohumeral capsular tensioning improves the proprioceptive capability of the shoulder and plays an important roll in restoring shoulder stability.

Several studies compared the proprioceptive capabilities of the shoulder between different surgical procedures, however only few have used the "dynamic unrestricted 3-dimensional arm movement model" that has been shown to be more appropriate for assessment of glenohumeral proprioception. To our knowledge, no previous study has compared proprioception measures of the glenohumeral joint following arthroscopic versus open repair for anterior shoulder instability, using the 3-dimensional unrestricted arm movement model.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least one year after a single operation for anterior shoulder instability of their dominant arm
* control subjects will be healthy volunteers with no history of shoulder complaints selected to match the age and gender of subjects

Exclusion Criteria:

* Neurological impairment involving the upper extremities
* Instability or recurrent dislocation of the operated shoulder
* Another surgery of the dominant extremity besides the single stabilization procedure

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients treated in our shoulder outpatients clinic will be candidates for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of smoothness parameters of subjects' shoulder movements. | At least 1 year following surgical repair for anterior shoulder instability

CONTACTS AND LOCATIONS:
Overall Officials: Dario Liebermann, PhD., Study Director — Department of Physical Therapy, Sackler Faculty of Medicine, Tel Aviv University, Israel; Moshe Peri (Pritsch), M.D, Study Chair — The Shoulder Surgery Unit, Sheba Medical Center, Tel Aviv University, Israel
Locations (1):
- Department of Physical Therapy, Sackler Faculty of Medicine, Tel Aviv University, Israel, Tel Aviv, Israel

REFERENCES:
- [Derived] Uri O, Pritsch M, Oran A, Liebermann DG. Upper limb kinematics after arthroscopic and open shoulder stabilization. J Shoulder Elbow Surg. 2015 Mar;24(3):399-406. doi: 10.1016/j.jse.2014.08.006. Epub 2014 Oct 22. PMID 25441562